CLINICAL TRIAL: NCT04696874
Title: Spectrum of Epididymis and Vas Deferens Anomalies Among Children With Cryptorchidism: A Retrospective Multi-center Study
Brief Title: Spectrum of Epididymis and Vas Deferens Anomalies Among Children With Cryptorchidism
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Magdy, Principle investigator, Aswan University Hospital
Other Study IDs: AswanUH1
Record Dates: First submitted 2020-12-18; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Epididymal Cyst; Vas Deferens; Anomaly
Keywords: epididymal cyst; duplicated vas deferens.; curled vas deferens; vanished testis
MeSH Terms: conditions — Spermatocele; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure:  — All testes were fixed to the ipsilateral sub-dartos pouch. All epididymides and vasa deferentia were carefully examined, and any observed anomalies were recorded.

SUMMARY:
: Data was collected retrospectively from six centers providing care for patients with undescended testicles from September 2017 to February 2019. All patients whose congenital anomalies of the epididymis or vas deferens were discovered incidentally during operative intervention for cryptorchidism and where photographs of the anomalies were taken were included.

DETAILED DESCRIPTION:
Background: Epididymal and vas deferens anomalies are not rare among children with cryptorchidism. They may affect fertility following orchiopexy.

Material and Methods: Data was collected retrospectively from six centers providing care for patients with undescended testicles from September 2017 to February 2019. All patients whose congenital anomalies of the epididymis or vas deferens were discovered incidentally during operative intervention for cryptorchidism and where photographs of the anomalies were taken were included.

ELIGIBILITY:
Inclusion Criteria:

- All included cases had photographic documentation.

Exclusion Criteria:

* cases without photographic documentation.

Ages: 8 Months to 125 Weeks | Sex: Male
Age Groups: Child
Study Population: We retrospectively collected data from patients with anomalies of the epididymis or vas deferens. These anomalies were discovered incidentally during operative intervention for cryptorchidism
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
collection of cases | one and half year
  retrospective from multicenter university hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Abdelmohsen, MD, Principal Investigator — Aswan University
Locations (1):
- Sarah Magdy Abdelmohsen, Cairo, P.O.Pox. 11331, Egypt

IPD SHARING:
Plan to Share IPD: Undecided